CLINICAL TRIAL: NCT00536822
Title: Prospective Assessment of Antioxidant Status of Pediatric Patients During Burn Rehabilitation
Brief Title: Antioxidant Status During Burn Rehabilitation
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn due to hospital emphasis on funded studies.
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michele Gottschlich, Research Scientist, Shriners Hospitals for Children
Other Study IDs: 07-06-04-01
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Burns
Keywords: rehabilitation; pediatrics
MeSH Terms: conditions — Burns

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — No specimens.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is believed that children with a prior history of significant burn injury continue to manifest low levels of antioxidants well into their convalescence.The purpose of this study is to examine malondialdehyde (an oxidative lipid marker) and vitamins E, C and beta carotene status in reconstructive burn patients.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 3 but less than 19 years
* Reconstructive or followup outpatient care at least 1 year postburn
* Initial burn size > 40%
* Written informed consent and HIPAA authorization

Exclusion Criteria:

* History of multivitamin or steroid use, liver disease, preburn malnutrition

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric burn
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
serum antioxidant levels | > 2 years postburn

CONTACTS AND LOCATIONS:
Overall Officials: Michele M Gottschlich, Principal Investigator — Shriners Hospital for Children